CLINICAL TRIAL: NCT05214456
Title: To Compare the Effect of Dry Needling Versus Lumbar Spine Mobilization on Symptoms in Patients With Chronic Nonspecific Low Back Pain
Brief Title: The Effect of Dry Needling Compared to Lumbar Spine Mobilization in Patients With Chronic Non Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR. IUMS.REC.1400.651
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain, dry needling, mobilization, pain pressure threshold, muscle function
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group will comprise 28 participants with chronic non-specific low back pain. The treatments of this group will include dry needling plus sham mobilization for the lumbar spine and routine physiotherapy. The needles will be inserted to obtain local twitch responses, and this process will continue until no more local twitch response occurs in each session. Then the needles will be left in place for 20 minutes. Sham mobilization for the lumbar spine will be done in the same way as the real mobilization, with the difference that the mobilization will be applied only on the skin surface and less than the first degree of Maitland's mobilization. Routine physical therapy will include low-level laser therapy and motor control training. The treatment will last 4 weeks, 8 sessions, twice a week.
  Interventions: Other: Dry needling
- Control group (Active Comparator): The control group will comprise 28 participants with chronic non-specific low back pain. The treatments of this group will include anterior-posterior mobilization based on the Maitland technique for the lumbar spine plus sham dry needling and routine physiotherapy. Based on the findings of the patient evaluation, the severity, rhythm, time, the degree of mobilization and the place of force (spine or lamina) will be determined. For sham dry needling The needles will be inserted subcutaneously and there will be no local twitch response. Then the needles will be left in place for 20 minutes. Routine physical therapy will include low-level laser therapy and motor control training. The treatment will last 4 weeks, 8 sessions, twice a week.
  Interventions: Other: Mobilization

INTERVENTIONS:
Other: Dry needling — The method of performing the dry needling technique will be based on the method presented by Dommerholt and Fernandez-de-las-Penas. The length of the needle (Tony, china) for each patient will be selected based on the size of the patient: 1) Multifidus: the patient will be placed in a prone position with a pillow under their belly to accommodate lumbar lordosis. The needles will be inserted into the lumbar multifidus muscles, 1.5 to 2 cm lateral to the spinous process of all lumbar vertebrates, perpendicular to the lamina (after piercing the skin, needles are directed inferomedially). 2) Quadratus lumborum: The patient will be placed in the side lying position with the side to be treated facing up. After identifying the lateral border of the quadratus lumborum muscle, the needle will be aimed straight downward in the direction of the transverse process, followed by slight anterior, posterior, and caudal needling to explore the entire muscle.
  Arms: Interventional group
Other: Mobilization — To perform Maitland's mobilization for lumbar spine, the anterior-posterior mobilization technique will be used and it is performed by pushing the heel (pisiform grip) or thumbs (thumb grip) to the vertebrae and can immediately reduce pain and restore motor function. First, the complete physical orthopedic evaluation of manual therapies will be performed using the Maitland evaluation method. Then, based on the findings of the patient evaluation, the severity, rhythm, duration and the degree of the mobilization and the place of force (spine or lamina) will be determined. To apply mobilization, the person will sleep in a prone position and the physiotherapist will use the heel of the hand or the thumbs to apply force to the first to fifth vertebrae of the lumbar spine. In segments that do not have a problem based on evaluation, first grade of the anterior-posterior Maitland's mobilization will be applied to the spinous process of the segment.
  Other Names: Non-thrust manipulation
  Arms: Control group

SUMMARY:
Low back pain is a major public health challenge worldwide. The aim of this study will be to compare the effect of dry needling with mobilization on pain, functional disability, quadratus lumborum and lumbar multifidus function, lumbar range of motion and pain pressure threshold using a randomized controlled trial design. pain and functional disability are primary outcomes and quadratus lumborum and lumbar multifidus function, lumbar range of motion and pain pressure threshold are considered as secondary outcomes. Patients will be randomly divided into two groups: The experimental group (dry needling, sham mobilization and routine physiotherapy) and the control group (mobilization, sham dry needling and routine physiotherapy).

DETAILED DESCRIPTION:
The present study will be a randomized, parallel group, two-arm, double-blind, double-dummy, superiority, controlled trial with a 1:1 allocation ratio. The main objective of this study is to compare the effects of dry needling and lumbar spinal mobilization on pain intensity, functional disability, lumbar multifidus and quadratus lumborum muscles function, lumbar range of motion and pain pressure threshold in patients with chronic non-specific low back pain. After selecting individuals with chronic non-specific low back pain by non-probability purposive sampling method, patients will be randomly assigned to two groups of dry needling (for lumbar Multifidus and Quadratus lumborum muscles) plus sham mobilization (first group) and lumbar spine mobilization plus sham dry needling group (second group). In addition, participants in both treatment groups will receive routine physiotherapy (including low-power laser and core stability exercise). Both groups will be treated for 8 sessions over 4 weeks. Primary outcomes include pain and functional disability, and secondary outcomes include quadratus lumborum and lumbar multifidus function, lumbar range of motion and pain pressure threshold. This study is a double-blind study in which the participants, the person evaluating the outcome, and the person analyzing the data will be blinded to the allocation of patients to the two treatment groups. All of the participants will be identified and recruited by posters and word-of-mouth from the university and the surrounding local communities. Eligible participants will be explained about the aim of the study and the examination involved in this study, and all eligible patients will sign a written informed consent before entering the study. The study will be performed in the Rehabilitation Sciences school of Iran University of Medical Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 to 45 years.
* Moderate pain intensity (between 30 to 60) based on Numerical Pain Rating Scale (0 means no pain and 100 is the most imaginable pain).
* Participants with trigger points in the quadratus lumborum and lumbar multifidus muscles.
* The Participant's symptoms are provoked with passive accessory intervertebral movements on at least one level of the lumbar spine vertebrae.
* Patients are able to read and write Persian.

Exclusion Criteria:

* Complications that affect the treatment process such as systemic diseases, neurological disorders, inflammatory conditions, infectious conditions, structural and degenerative changes, metabolic bone diseases and bleeding disorders.
* History of lumbar surgery.
* Specific low back pain (Neurogenic low back pain, spinal stenosis, cauda equina syndrome, spondylolisthesis, and Presence of any signs or symptoms of non- musculoskeletal pathology e.g. cancer, infection and fracture based on paraclinical findings)
* Inability to obtain prone lying.
* Pregnancy.
* Needle phobia.
* Long history of steroid use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Pain intensity measurement before intervention and 7 days after intervention
  Mean Change from Baseline in Pain Scores on the Numerical Pain Rating Scale (0 means no pain and 100 means the most imaginable pain).
  9
Functional disability | Before intervention and 7 days after intervention
  Mean Change from Baseline in Functional disability Scores based on Oswestry Disability Index. 0% to 20% indicate minimal disability, 21% to 40% indicate moderate disability, 41%-60% indicates severe disability, 61%-80% means crippled and 81%-100% indicates that the patient is either bed-bound or exaggerating his/her symptoms. The validity and the reliability of the Persian version of this questionnaire has been shown in the previous studies.

SECONDARY OUTCOMES:
Lumbar multifidus and quadratus lumborum muscles functional change | Before intervention and 7 days after intervention
  Mean Change from Baseline in Lumbar multifidus and quadratus lumborum muscles Functional changes based on the measurement of thickness changes between rest and contraction status of these muscles by using ultrasound.
Range of motion | Before intervention and 7 days after intervention
  Mean Change from Baseline in Range of motion based on the measurement with tape
Pain pressure threshold | Before intervention and 7 days after intervention
  Mean Change from Baseline in Pain pressure threshold based on measurement with algometer

CONTACTS AND LOCATIONS:
Overall Officials: Hamide Mirzaie, MSc student, Principal Investigator — Iran University of Medical Sciences; Mohammadreza Pourahmadi, PhD, Study Director — Iran University of Medical Sciences
Locations (1):
- IRANums, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available on a reasonable request to the corresponding author.
Supporting Information: Study Protocol
Time Frame: starting 6 months after the publication
Access Criteria: The data will be available for physical therapists working in academic institutions and also clinicians working in the field of musculoskeletal disorders. The raw data and results of this study can be used in future relevant systematic reviews. Thus, the raw data and results of this study will be available for researchers working in the field of low back pain. Applicants can contact hamide mirzaie by Email. Email address: hamide.mirzaie@yahoo.com. Applicants should explain their project and how the data/documents of this study will be used in their project in detail. Then, the data/documents files will be sent by email to applicants on request. This process may takes 10-12 working days.

REFERENCES:
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Coulter ID, Crawford C, Hurwitz EL, Vernon H, Khorsan R, Suttorp Booth M, Herman PM. Manipulation and mobilization for treating chronic low back pain: a systematic review and meta-analysis. Spine J. 2018 May;18(5):866-879. doi: 10.1016/j.spinee.2018.01.013. Epub 2018 Jan 31. PMID 29371112
- [Background] Couto C, de Souza IC, Torres IL, Fregni F, Caumo W. Paraspinal stimulation combined with trigger point needling and needle rotation for the treatment of myofascial pain: a randomized sham-controlled clinical trial. Clin J Pain. 2014 Mar;30(3):214-23. doi: 10.1097/AJP.0b013e3182934b8d. PMID 23629597
- [Background] Dommerholt J, Fernández-de-las-Peñas C. Trigger point dry needling e-book: an evidence and clinical-based approach: Elsevier Health Sciences; 2018.
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] Itoh K, Katsumi Y, Hirota S, Kitakoji H. Effects of trigger point acupuncture on chronic low back pain in elderly patients--a sham-controlled randomised trial. Acupunct Med. 2006 Mar;24(1):5-12. doi: 10.1136/aim.24.1.5. PMID 16618043
- [Background] Thiry P, Reumont F, Brismee JM, Dierick F. Short-term increase in discs' apparent diffusion is associated with pain and mobility improvements after spinal mobilization for low back pain. Sci Rep. 2018 May 29;8(1):8281. doi: 10.1038/s41598-018-26697-7. PMID 29844484
- [Background] Pecos-Martin D, de Melo Aroeira AE, Veras Silva RL, Martinez de Tejada Pozo G, Rodriguez Solano LM, Plaza-Manzano G, Gallego-Izquierdo T, Falla D. Immediate effects of thoracic spinal mobilisation on erector spinae muscle activity and pain in patients with thoracic spine pain: a preliminary randomised controlled trial. Physiotherapy. 2017 Mar;103(1):90-97. doi: 10.1016/j.physio.2015.10.016. Epub 2015 Dec 12. PMID 27012824
- [Background] Elly H. Maitland's vertebral manipulation, management of Neuromusculoskeletal disorders. London: Churchill Livingstone. 2013.
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Liu IS, Chai HM, Yang JL, Wang SF. Inter-session reliability of the measurement of the deep and superficial layer of lumbar multifidus in young asymptomatic people and patients with low back pain using ultrasonography. Man Ther. 2013 Dec;18(6):481-6. doi: 10.1016/j.math.2013.04.006. Epub 2013 May 28. PMID 23726537
- [Background] Schryver A, Rivaz H, Rizk A, Frenette S, Boily M, Fortin M. Ultrasonography of Lumbar Multifidus Muscle in University American Football Players. Med Sci Sports Exerc. 2020 Jul;52(7):1495-1501. doi: 10.1249/MSS.0000000000002292. PMID 32028457
- [Background] Fraeulin L, Holzgreve F, Brinkbaumer M, Dziuba A, Friebe D, Klemz S, Schmitt M, Theis A AL, Tenberg S, van Mark A, Maurer-Grubinger C, Ohlendorf D. Intra- and inter-rater reliability of joint range of motion tests using tape measure, digital inclinometer and inertial motion capturing. PLoS One. 2020 Dec 10;15(12):e0243646. doi: 10.1371/journal.pone.0243646. eCollection 2020. PMID 33301541
- [Background] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Background] Pourahmadi MR, Ebrahimi Takamjani I, Jaberzadeh S, Sarrafzadeh J, Sanjari MA, Mohsenifar H, Bagheri R, Taghipour M. The Effect of Core Stabilization Exercise on the Kinematics and Joint Coordination of the Lumbar Spine and Hip During Sit-to-Stand and Stand-to-Sit in Patients With Chronic Nonspecific Low Back Pain (COSCIOUS): Study Protocol for a Randomized Double-Blind Controlled Trial. JMIR Res Protoc. 2017 Jun 1;6(6):e109. doi: 10.2196/resprot.7378. PMID 28572078
- [Background] Pourahmadi MR, Bagheri R, Jannati E, Ebrahimi Takamjani I, Sarrafzadeh J, Mohsenifar H. Effect of Elastic Therapeutic Taping on Abdominal Muscle Endurance in Patients With Chronic Nonspecific Low Back Pain: A Randomized, Controlled, Single-Blind, Crossover Trial. J Manipulative Physiol Ther. 2018 Sep;41(7):609-620. doi: 10.1016/j.jmpt.2017.10.019. Epub 2018 Aug 8. PMID 30098819
- [Background] Clark BC, Russ DW, Nakazawa M, France CR, Walkowski S, Law TD, Applegate M, Mahato N, Lietkam S, Odenthal J, Corcos D, Hain S, Sindelar B, Ploutz-Snyder RJ, Thomas JS. A randomized control trial to determine the effectiveness and physiological effects of spinal manipulation and spinal mobilization compared to each other and a sham condition in patients with chronic low back pain: Study protocol for The RELIEF Study. Contemp Clin Trials. 2018 Jul;70:41-52. doi: 10.1016/j.cct.2018.05.012. Epub 2018 May 21. PMID 29792940
- [Background] Wang-Price S, Zafereo J, Couch Z, Brizzolara K, Heins T, Smith L. Short-term effects of two deep dry needling techniques on pressure pain thresholds and electromyographic amplitude of the lumbosacral multifidus in patients with low back pain - a randomized clinical trial. J Man Manip Ther. 2020 Dec;28(5):254-265. doi: 10.1080/10669817.2020.1714165. Epub 2020 Jan 17. PMID 31960773
- [Background] Benito-de-Pedro M, Becerro-de-Bengoa-Vallejo R, Elena Losa-Iglesias M, Rodriguez-Sanz D, Lopez-Lopez D, Palomo-Lopez P, Mazoteras-Pardo V, Calvo-Lobo AC. Effectiveness of Deep Dry Needling vs Ischemic Compression in the Latent Myofascial Trigger Points of the Shortened Triceps Surae from Triathletes on Ankle Dorsiflexion, Dynamic, and Static Plantar Pressure Distribution: A Clinical Trial. Pain Med. 2020 Feb 1;21(2):e172-e181. doi: 10.1093/pm/pnz222. PMID 31502640
- [Background] Griswold D, Gargano F, Learman KE. A randomized clinical trial comparing non-thrust manipulation with segmental and distal dry needling on pain, disability, and rate of recovery for patients with non-specific low back pain. J Man Manip Ther. 2019 Jul;27(3):141-151. doi: 10.1080/10669817.2019.1574389. Epub 2019 Feb 9. PMID 30935327
- [Derived] Mirzaei Ashani H, Pourahmadi M, Ayoubpour MR, Dadgoo M, Sarrafzadeh J, Firouze B. The Effect of Dry Needling Compared to Lumbar Spine Mobilization on Functional Disability in Patients with Nonspecific Chronic Low Back Pain: Study Protocol for a Randomized Controlled Trial. Adv Biomed Res. 2025 Aug 26;14:80. doi: 10.4103/abr.abr_318_23. eCollection 2025. PMID 40958926